CLINICAL TRIAL: NCT01522105
Title: Evaluation of Cerebrospinal Fluid Concentration of Daptomycin (Cubicin¬) in Pediatric Patients With Gram-positive Bacterial Meningitis, Concurrently Receiving Standard Antimicrobial Therapy
Brief Title: Daptomycin in Pediatric Patients With Bacterial Meningitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient patient recruitment
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 046/11; 2012DR1007 (Other: Swissmedic); 2049
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Meningitis
Keywords: Meningitis; Central Nervous System Infections; Pediatrics; Daptomycin; Anti-Bacterial Agents; Therapeutic Use; Pharmacologic Actions
MeSH Terms: conditions — Meningitis; Central Nervous System Infections | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): i.v. daptomycin given 24 hours after first ceftriaxone dose at age appropriate dosage
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — One dose of daptomycin given at an age appropriate dosage (3-24 months 6mg/kg; 2-6 years 10mg/kg; 7-11 years 8mg/kg; 12-16years 6mg/kg)

SUMMARY:
5 Children > 3months and < 16 years with Gram-positive meningitis will receive a single dose of daptomycin 24 hours after the first dose of ceftriaxone. 4-8 hours after daptomycin administration a second lumbar puncture is performed to determine the peak concentration of daptomycin in the cerebrospinal fluid. In parallel peak and trough level of daptomycin will be measured in the plasma. The investigators anticipate that daptomycin penetrates into the cerebrospinal fluid in bactericidal concentrations

DETAILED DESCRIPTION:
Background

Acute bacterial meningitis is a severe infection, which leads to persistent neurological deficits in up to 50% of patients, despite optimal medical treatment. Although, the incidence of acute bacterial meningitis has declined in developed countries since the advent of vaccines against Haemophilus influenzae and Streptococcus pneumoniae, this is not yet true for developing countries. Also, the impact of serotype replacement in invasive pneumococcal disease cannot be estimated to date.

Acute bacterial meningitis causes brain injury most prominently in the cerebral cortex, the inner ear and in the hippocampus. In the hippocampus, a brain region functionally important for learning and memory, the brain damage is characterized by apoptosis of cells in the hippocampal dentate gyrus. Autopsy studies demonstrated the occurrence of apoptosis in neurons of the hippocampal dentate gyrus in the majority (> 75%) of human autopsy cases, who died of acute bacterial meningitis. Children are particularly vulnerable to this form of brain damage because of ongoing development of neurological functions and they have a higher risk of neurologic deficits after bacterial meningitis than adults. The 3 most common pathogens in childhood meningitis are Streptococcus pneumoniae, Haemophilus influenzae and Neisseria meningitidis. Streptococcus pneumoniae is associated with the greatest risk for fatal outcome or persistent neurological deficits. In the most recent prospective study hearing loss was the most common major sequelae in half of the patients, followed by cognitive deficits (40.0%), seizures (21.2%), and motor deficits (21.2%); one third of these patients had multiple defects.The pathogenesis of brain damage in meningitis is driven by the host's owns inflammatory reaction to the invading pathogens in the subarachnoid space. This inflammatory reaction is triggered by the release of subcapsular bacterial components. Unfortunately, β-lactam antibiotics, current standard of care in bacterial meningitis, induce bacteriolysis leading to a brisk accumulation of subcapsular bacterial components in the cerebrospinal fluid (CSF), which in turn trigger an over-shooting inflammatory reaction contributing to brain damage.

First evaluated more than 50 years ago, adjunctive corticosteroids still are the only approved therapy to minimize this inflammatory reaction in humans.

In children the benefit of a combination therapy with dexamethasone and ceftriaxone has only been proven in the reduction of permanent hearing loss after Haemophilus influenzae type b meningitis, a pathogen that today is virtually eradicated in regions that implemented the vaccination. Furthermore, the beneficial effects of dexamethasone administration in meningitis have been challenged repeatedly. A recent prospective study and two meta-analyses show conflicting results considering the benefit of adjuvant corticosteroid treatment for neurological outcome in children with acute bacterial meningitis. Furthermore, adjunctive corticosteroid treatment does not seem to benefit patients with acute bacterial meningitis in developing countries. Even more worrying are results in experimental meningitis, which indicate that dexamethasone might lead to neuronal injury.

Daptomycin (Cubicin¨, Novartis Pharma AG, Basel Switzerland) is a cyclic lipopeptide antimicrobial agent active against most Gram-positive bacteria including strains that are resistant to methicillin, vancomycin or linezolid. It binds to the membrane of Gram-positive bacteria and causes rapid depolarization of membrane potential leading to bacterial cell death. Thereby, daptomycin exerts a bactericidal, but non-bacteriolytic effect and does not cause release of subcapsular bacterial components.

Recently, it has been proven for experimental pneumococcal meningitis that daptomycin leads to a substantially reduced inflammatory reaction compared to ceftriaxone. Additionally, it has been shown that compared to ceftriaxone monotherapy, daptomycin plus ceftriaxone lowers the levels of pro-inflammatory mediators in the cerebrospinal fluid (CSF) and reduces brain damage in the form of hippocampal apoptosis and hearing loss in infant rat pneumococcal meningitis.

Based on the experimental data summarized above, it appears reasonable to assume that the use of daptomycin, followed by the administration of a broad-spectrum antimicrobial agent in children with pneumococcal meningitis, or other Gram-positive meningitis, would lead to a reduced inflammatory response and, ultimately, to a reduced incidence of permanent neurological deficits.

While it has been established that the pharmacokinetics (PK) of daptomycin in children are age-dependent 6, only scarce data exist on the extent of penetration of daptomycin into the inflamed CSF. Anecdotal evidence indicates that in humans with inflamed meninges daptomycin penetrates into the CSF in sufficient amounts. This is supported by animal studies.

There are currently two pediatric studies ongoing in the United States of America. DAP-PEDS- 09-01 will assess pharmacokinetics (PK) and safety of Daptomycin in 18 children ages 3-24 months with Gram-positive bacterial infections. DAP-PEDS-07-03 will assess efficacy and safety of multiple daptomycin doses in 339 children aged 2 - 17 years with skin and skin structures infections. Design and dosing of both studies are based on previous findings in two pediatric studies involving 25 children ages 2-17 years and 12 children ages 2-6 years. None of these studies will or has investigated daptomycin penetration into the CSF.

As a first step to establishing optimal dosing recommendations for daptomycin in pediatric patients with meningitis, the present pharmacokinetic study attempts to document adequate CSF penetration of daptomycin in children with acute bacterial meningitis.

Objective

Characterize the extent to which daptomycin penetrates into the CSF of children with acute bacterial meningitis. Because determination of AUC in the CSF is not feasible, Cmax of daptomycin in the CSF will be taken as a surrogate marker

Methods

Children between the ages of 3 months to 16 years with acute bacterial meningitis will be recruited. After obtaining baseline blood parameters including muscular enzymes, renal function, hepatic function, and blood cultures, a lumbar puncture is performed and standard of care therapy with ceftriaxone 100mg/kg (top dose 4g i.v.) is initiated. 24 hours after hospitalisation a single dose of daptomycin at an age- dependent dosage, is administered i.v. over 15 min. shortly before or after the second dose of ceftriaxone. 4-8 hours after daptomycin administration a second lumbar puncture is performed to obtain a CSF sample for measurement of peak daptomycin levels. Serum concentrations of daptomycin are measured immediately after i.v. administration, at the time of lumbar puncture and 24 hours after daptomycin administration.

Daptomycin therapy is discontinued after one dose, while standard of care antimicrobial therapy is continued for a total of 7 to 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Age > 3 months and < 16 years
* Bacterial meningitis
* Written parental (or appropriate legal representative) informed consent prior to study inclusion

Exclusion Criteria

* Gram-negative bacteria in the CSF
* Creatinine clearance < 80ml/min/1.73m2
* Creatinine phosphokinase level > 2x upper age related norm
* Known allergy or hypersensitivity to daptomycin
* Known clinical significant cardiovascular, pulmonary, renal, hepatic, gastrointestinal, endocrine, hematologic, autoimmune disease, or primary immunodeficiency
* Height and weight below 3rd or above 95th percentile
* History of, or current muscular disease
* Underlying neurological disease with disruption of blood brain barrier
* Epilepsy
* Muscular weakness, history of peripheral neuropathy, or Guillain-Barré syndrome

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Characterization of the peak concentration of daptomycin in the cerebrospinal fluid of pediatric patients with bacterial meningitis | 4-8 hours after drug administration

SECONDARY OUTCOMES:
Evaluate possible side effects of daptomycin in pediatric patients with bacterial meningitis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Agyeman, MD, Principal Investigator — University Children's Hospital Bern
Locations (1):
- Dep. of Pediatrics, University Hospital Bern, Bern, Switzerland